CLINICAL TRIAL: NCT03973359
Title: Incidence, Outcome and Prevention of Congenital Human Cytomegalovirus (HCMV) Infection in HCMV-seropositive Pregnant Women
Brief Title: Epidemiology and Prevention of Congenital HCMV in Immune Mothers. Congenital HCMV Infection Lombardy
Acronym: CHILd
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Fondazione Regionale per la Ricerca Biomedica (Other)
Responsible Party: Principal Investigator, Daniele Lilleri, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20170011101
Record Dates: First submitted 2019-05-20; First posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Congenital Cytomegalovirus Infection; Maternal Cytomegalovirus Infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidemiology (No Intervention): HCMV-seropositive pregnant women receiving standard care
- Prevention (Experimental): HCMV-seropositive pregnant women receiving hygienic information
  Interventions: Behavioral: Hygienic recommendations

INTERVENTIONS:
Behavioral: Hygienic recommendations — Recommendation of protective behaviours such as frequent hand washing and avoiding risky behaviours such as kissing young children on the mouth or cheeks and sharing utensils, foods etc.
  Arms: Prevention

SUMMARY:
Human cytomegalovirus (HCMV) is the leading infectious agent causing congenital disabilities such as mental retardation, psychomotor delay, hearing loss, speech and language disabilities, behavioural disorders and visual impairment. About 0.6% newborns are HCMV-congenitally infected and, among these, about 20% are symptomatic at birth or will develop long-term sequelae. The public health impact of congenital HCMV is substantial although greatly unrecognized. In Italy, estimated direct costs per affected child exceed €100.000 for a total of €60-70M. HCMV is also a significant cause of infection/disease in the immunocompromised host.

Epidemiological studies and population-based models have preliminarily documented that most of the burden associated to congenital HCMV would be due to non-primary maternal infection. Presently, reinfections are believed to be responsible for the great majority of infected fetuses born to immune mothers.

This study addresses incidence, outcome and prevention of congenital HCMV infection in seropositive pregnant women.The study includes 2 parts: part 1 in which the incidence and outcome of congenital HCMV is investigated in a large population of HCMV seropositive pregnant women and HCMV shedding and immune response is closely monitored in a subset of participants (nested study); part 2 in which the efficacy of an hygiene intervention is assessed.

DETAILED DESCRIPTION:
Part 1. Epidemiologic study. To investigate incidence and outcome of congenital infection in immune mothers, clinical records of pregnant women are reviewed for HCMV serostatus at ≤ 13 weeks' gestation. Women with HCMV serology compatible with a remote infection are asked to participate in the study. Consenting women are given a pre-stamped, pre-addressed envelope containing a swab to collect newborn's saliva. Envelopes are sent by courier to a centralized diagnostic facility for HCMV testing.

Women can also be enrolled at delivery, provided that the woman has records of presence of virus-specific IgG and absence of IgM early during gestation(or in a previous pregnancy) or, in case of unknown serostatus, a sample of serum/plasma stored at ≤ 13 weeks' gestation is available for retrospective antibody testing (retrospective part of the epidemiology study).

Part 1. Nested study. A subset of IgG pos IgM neg women selected among those enrolled at ≤13 weeks' gestation in the epidemiology study are included in a nested study. These women are monitored at enrolment, 20, 30 weeks of gestation and at delivery by prospective determination of HCMV DNA excretion in different bodily fluids. In DNA-positive specimens selected HCMV genes will be sequenced.

Part 2. Prevention study. To assess the effectiveness of hygiene measures for prevention of congenital infection HCMV seropositive pregnant women are enrolled at ≤ 13 weeks' gestation. Part 2 starts when enrolment of Part 1 is completed. In practice, part 2 is a continuation of part 1 with the only addition of delivering hygiene information at enrolment.

Part 2 will not be performed in case congenital infection rate in Part 1 is <0.4% and clear maternal risk factor for intrauterine transmission cannot be identified at interim analysis (i.e. after examination of 5000 newborns).

In case HCMV DNA is detected in newborn's saliva, a urine sample is obtained for confirmation of congenital infection. Infants with documented congenital infection are clinically assessed at the time of diagnosis (for Part 1 and 2) and at one year of age (Part 1 only).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old) pregnant women at ≤13 weeks gestation
* Presence of HCMV IgG and absence of IgM or presence of high avidity IgG with or without IgM
* Presence of HCMV-specific IgG and absence of IgM or presence of high avidity IgG in case of positive IgM at ≤13 weeks gestation documented by medical report or by retrospective antibody determination on samples stored at ≤13 weeks (for women enrolled at delivery)
* Willingness to participate in the study
* Ability to understand information material
* Written informed consent

Exclusion Criteria:

* Unreliable women as judged by the investigator
* Women not willing to give written consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23500 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Part 1. Epidemiology study. Incidence and clinical outcome of congenital HCMV infection in pregnant women with preconception immunity. | Within 21 days of life
  Number of infants with ascertained congenital infection.
Part 2. Prevention study. Efficacy of hygiene counseling in reducing congenital HCMV infection in pregnant women with preconception immunity. | Within 21 days of life
  Number of infants with ascertained congenital infection born to HCMV seropositive women informed about hygiene measures compared to the number of newborns with congenital infection diagnosed in Part 1.

SECONDARY OUTCOMES:
Frequency of non-primary infections during pregnancy (Nested study) | 10, 20, 30, 40 gestation weeks
  Number of participants with HCMV non-primary infection. HCMV non-primary infection is defined as detection of HCMV DNA shedding in bodily fluids.
Frequency of HCMV re-infections vs re-activations during pregnancy (Nested study) | 10, 20, 30, 40 gestation weeks
  Number of participants with HCMV re-infection or re-activation. Re-infection is defined as the appearance of genetically distinct HCMV strains; Reactivation is defined as the sustained presence of the same strain.
Antigen-specific IgG levels in non-primary infection during pregnancy (Nested study) | 10, 20, 30, 40 gestation weeks
  Levels of antigen-specific IgG in participants with or w/o non-primary infection.
Antigen-specific IgM levels in non-primary infection during pregnancy (Nested study) | 10, 20, 30, 40 gestation weeks
  Levels of antigen-specific IgM in participants with or w/o non-primary infection.
Neutralizing antibody titers in non-primary infection during pregnancy (Nested study) | 10, 20, 30, 40 gestation weeks
  Titers of neutralizing antibodies in participants with or w/o non-primary infection.
Risk factors for congenital HCMV infection in pregnant women with preconception immunity. Age | Delivery
  Age in mothers of newborns with or w/o congenital HCMV infection
Risk factors for congenital HCMV infection in pregnant women with preconception immunity. Country of origin | Delivery
  Country of origin of mothers of newborns with or w/o congenital HCMV infection
Risk factors for congenital HCMV infection in pregnant women with preconception immunity. Occupation | Delivery
  Occupation of mothers of newborns with or w/o congenital HCM infection
Risk factors for congenital HCMV infection in pregnant women with preconception immunity. Contact with young children | Delivery
  Contact with children <36 months in mothers of newborns with or w/o congenital HCMV infection
Risk factors for congenital HCMV infection in pregnant women with preconception immunity. Twin pregnancy | Delivery
  Twin vs singleton pregnancy in mothers of newborns with or w/o congenital HCMV infection
Risk factors for congenital HCMV infection in pregnant women with preconception immunity. Concomitant pathologies | Delivery
  Concomitant pathologies in mothers of newborns with or w/o congenital HCMV infection

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Lilleri, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (12):
- Italy (12):
  - ASST Spedali Civili di Brescia, Brescia
  - Poliambulanza Brescia, Brescia
  - ASST Vimercate (Ospedale di Carate Brianza), Carate Brianza
  - ASST Monza (presidio di Desio), Desio
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Milan
  - Ospedale Macedonio Melloni (ASST FBF-Sacco), Milan
  - Ospedale San Raffaele, Milan
  - Ospedale Buzzi (ASST FBF-Sacco), Milan
  - Ospedale Sacco (ASST FBF-Sacco), Milan
  - Fondazione Monza Brianza per il Bambino e la sua Mamma, Monza
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - ASST dei Sette Laghi (Ospedale Filippo Del Ponte), Varese

REFERENCES:
- [Derived] Lilleri D, Tassis B, Pugni L, Ronchi A, Pietrasanta C, Spinillo A, Arossa A, Achille C, Vergani P, Ornaghi S, Riboni S, Cavoretto P, Candiani M, Gaeta G, Prefumo F, Fratelli N, Fichera A, Vignali M, Barbasetti Di Prun A, Fabbri E, Cetin I, Locatelli A, Consonni S, Rutolo S, Miotto E, Savasi V, Di Giminiani M, Cromi A, Binda S, Fiorina L, Furione M, Cassinelli G, Klersy C; CHILd Study Group. Prevalence, Outcome, and Prevention of Congenital Cytomegalovirus Infection in Neonates Born to Women With Preconception Immunity (CHILd Study). Clin Infect Dis. 2023 Feb 8;76(3):513-520. doi: 10.1093/cid/ciac482. PMID 35717635